CLINICAL TRIAL: NCT06933225
Title: OPEN-LABEL STUDY TO EVALUATE THE SAFETY AND EFFICACY OF A MICRONEEDLING DEVICE USED IN FACIAL AESTHETICS
Brief Title: SAFETY AND EFFICACY OF A MICRONEEDLING DEVICE USED IN FACIAL AESTHETICS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Circa Skin Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22E1008; 2024-A01913-44 (Other: ANSM registration number)
Record Dates: First submitted 2025-04-08; First posted 2025-04-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WOW fusion Microneedling Device, 1.00 mm (Experimental): One treatment session on the whole face, on D0 and second treatment on D30.
  Interventions: Other: WOW fusion Microneedling Device, 1.00 mm

INTERVENTIONS:
Other: WOW fusion Microneedling Device, 1.00 mm — One treatment session on the whole face, on D0 and second treatment on D30.

SUMMARY:
Microneedling (MN), also referred to as collagen induction therapy, uses small needles to create mechanical injury to the skin. The basis of MN relies on physical trauma. It has been proposed that the trauma generated by needle penetration in the skin induces regeneration of the dermis The needles penetrate the stratum corneum and create small holes known as micro-conduits with minimal damage to the epidermis.

MN therapy is widely used to improve the appearance of facial scars, stretch marks and rejuvenate photoaged skin. Recently, it has been shown that MN can improve skin wrinkles on the face. MN can be used alone or to increase absorption of topical medications, growth factors, or deliver radiofrequency directly to the dermis.

The product tested is a microneedling device with 20 micro-needles of 1.00 mm depth penetration. This microneedling device is considered as a medical device in the US but not in Europe, according to Appendix XVI of the European regulation on medical devices 2017/745 of 5 April 2017. It is not yet commercialized neither in Europe nor in US. This first-in-man, pilot, clinical study is designed to first confirm the cutaneous tolerance of the device and provide some first data on device performance. For this purpose, 33 subjects with mild to moderate wrinkles on the face and seeking improvement of his/her face aspect, will be treated on Day 0 and Day 30 with the microneedling device on the face. Follow-up visits will be done 30 and 60 days after first treatment. Treatment Site Reactions (TSR) and Adverse reactions (ARs) will be collected to evaluate the device safety. Change from baseline of wrinkle severity and Global Aesthetic Improvement Scale (GAIS) will be used to evaluate product performance. Subject evaluation will also be analysed, and photos will be taken to illustrate device effect.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject.
2. Sex: male and female
3. Age: 18 years or older
4. Subject seeking an improvement of her/his face aspect using an aesthetic procedure.
5. Subject with mild to moderate wrinkles (grade 1, 2 or 3 on the 6-points Lemperle Scales) on at least 2 of the following area:

   * Horizontal forehead lines
   * Periorbital lines
   * Cheek folds
6. Subject willing to abstain from other facial aesthetic procedure in the full face through the entire study duration.
7. Subject having given their free, express, and informed consent.
8. Subject psychologically able to understand the information related to the study, and to give their written informed consent.
9. Subject registered with a social security scheme.
10. Female of childbearing potential must use a medically accepted contraceptive method since at least 12 weeks before the beginning of the study and throughout the study.
11. Female subjects of childbearing potential must have a negative pregnancy test at the inclusion.

Exclusion Criteria:

* 1. Subjects who are pregnant, nursing or intend to become pregnant during study participation.

  2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.

  3. Subject in a social or sanitary establishment. 4. Subjects that are currently enrolled in another drug or device study. 5. Subject with an excessive consumption of alcohol (more than 2 glasses of wine per day) and/or tobacco (more than 10 cigarettes per day).

  6. Subjects with a history of allergies or hypersensitivity to any components or ingredients in the device (especially allergy to nickel or gold).

  7. Subjects with severe allergies manifested by a history of anaphylaxis, or history or presence of multiple and severe allergies.

  8. Subjects that have any skin pathology or condition including tattooing or scarring that could interfere with the evaluation of the treatment areas.

  9. Subjects who suffer from rosacea, eczema, psoriasis, atopic dermatitis, sun-burned or broken skin, inflammatory or irritated skin conditions, active cold sores, moderate to severe acne, abscess, herpes, unhealed wound, cancerous or precancerous lesion on the face.or are taking any prescribed medication for their skin or any skin disease.

  10. Subject with any skin or systemic disease (acute and/or chronic), in the previous year, likely to interfere with the measured parameters or to put the subject to an undue risk.

  11. Subject with known history of or suffering from autoimmune disease and/or immune deficiency.

  12. Subject predisposed to keloids or hypertrophic scarring. 13. Subjects who have a hemorrhagic (bleeding) disorder or hemostatic (bleeding) dysfunction.

  14. Subject with pigmentation disorders (vitiligo, melasma,….). 15. Subjects who have had any form of collagen soft tissue treatment within the last 12 months.

  16. Subject having resorbable filling product (e.g., hyaluronic acid) injections, an ultrasound-based treatment, a dermabrasion, a deep chemical peeling or other ablative procedure on the face within the past 12 months prior to study start and a facial surgery in the past 2 years.

  17. Subject having received injections of permanent (e.g., acrylate polymers, silicone, polytetrafluoroethylene) or semi-permanent filling on the face (L Polylactic acid, Calcium Hydroxyapatite...).

  18. Subject with subcutaneous retaining structure on the face (meshing, threads, gold strand).

  19. Subjects having received botulinum toxin in the face within the 9 previous months.

  20. Subject having received mesotherapy products in the face within the 6 previous months.

  21. Subject having done a superficial or medium peeling or a superficial scrub on the face or having received LED or laser treatment on the face within the 2 previous months.

  22. Subject having used cosmetic products with alpha hydroxy acids (AHA) in the previous month.

  23. Subjects who are currently, or within the past 3 months, treated with any systemic immunosuppressive therapy including but not limited to chemotherapy agents or corticosteroids (including inhaled or insufflated corticosteroids).

  24. Subjects who are currently, or within the past 3 months, treated with any topical OTC drug or prescription therapy on their face.

  25. Subjects taking an antithrombotic, antiplatelet or other blood thinning medications in the past 3 months.

  26. Subject taking food supplement with an effect on skin quality (collagen, DHEA, …) in the 3 previous months.

  27. Subjects that have received an investigational drug or device within 30 days prior to entering this study.

  28. Subject receiving any treatment that, in the opinion of the clinical investigator, may interfere with test results or put the subject to undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Participant with treatment site reaction | 30 days after Day 0 and 30 days after Day 30
  evaluated on a scale from 0 (None) to 3 (Severe)

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale assessment (GAIS) | Day 30 and Day 60
  evaluated by the investigator. 5 point scale from 1 : very much improved to 5 worsening.
Global Aesthetic Improvement Scale assessment (GAIS) | Day 30 and Day 60
  evaluated by the subject. 5 point scale from 1 : very much improved to 5 worsening.
Lemperle Wrinkle Scales | Day 0, Day 30 and Day 60
  Evaluated by the investigator. 6 point scale as follow :
  0: No wrinkle
  1. Just perceptible wrinkles
  2. Shallow wrinkles
  3. Moderately deep wrinkles
  4. Deep wrinkles, well-defined edges
  5. Very deep wrinkles, redundant folds
Average roughness with fringe projection system | Day 30 and Day 60
  Average height of the roughness (average relief) = Rz Average roughness (average relief) = Ra Maximum height of the roughness (maximum relief amplitude) = Rz
  will be calculated direclty from fringe projection system software
Maximum height with fringe projection system | Day 30 and Day 60
Average height with fringe projection system | Day 30 and Day 60
Satisfaction of the injectors | Day 0 and Day 30
  Will be evaluated by a questionnaire on a 5 point scale : 1 very satisfied to 5 very dissatisfied
Satisfaction of the subject | Day 30 and Day 60
  Will be evaluated by a questionnaire on a 5 point scale : 1 very statisfied to 5 verry dissatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Pharmascan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No